CLINICAL TRIAL: NCT01139775
Title: A Phase 1/Randomized Phase 2 Study to Evaluate LY2603618 in Combination With Pemetrexed and Cisplatin in Patients With Stage IV Non-small Cell Lung Cancer
Brief Title: A Study in Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13797; I2I-MC-JMMG (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-06-01; First posted 2010-06-09 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: solid tumors; Mesothelioma; Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma; Carcinoma | interventions — Pemetrexed; Cisplatin; LY2603618

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1: LY2603618 130 to 275 mg (Experimental): Cycle 1-2 (21-day cycle):
  Day 1: pemetrexed 500 milligrams per meter square (mg/m^2) + cisplatin 75 mg/m^2
  Day 2: LY2603618 at 130-275 milligrams (mg)
  After 2 cycles, participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion is met.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: LY2603618
- Phase 2: Pemetrexed + Cisplatin + LY2603618 (Experimental): Cycles 1-4 (21-day cycle):
  Before 25 Oct 2012:
  Day 1: pemetrexed 500 mg/m^2 + cisplatin 75 mg/m^2
  Day 2: LY2603618 dose from phase 1 portion of trial
  After 25 Oct 2012:
  Day 1: pemetrexed 500 mg/m^2 + cisplatin 75 mg/m^2
  After 4 cycles, participants may continue on maintenance therapy until disease progression, unacceptable toxicity, or other withdrawal criterion is met.
  Maintenance Therapy Experimental Arm (every 21 days):
  Before 25 Oct 2012:
  Day 1: pemetrexed 500 mg/m^2
  Day 2: LY2603618 dose determined from phase 1
  After 25 Oct 2012:
  Day 1: pemetrexed 500 mg/m^2
  If, as of 25 Oct 2012, participant was in maintenance therapy and randomized to the experimental arm, the participant is eligible to continue with pemetrexed (Day 1)/LY2603618 (Day 2) therapy if the investigator deems it is in the best interest of the participant and the participant consents.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: LY2603618
- Phase 2: Pemetrexed + Cisplatin (Active Comparator): Cycle 1-4 (21-day cycle):
  Day 1: pemetrexed 500 mg/m^2 + cisplatin 75 mg/m^2
  After 4 cycles, participants may continue on maintenance therapy until disease progression, unacceptable toxicity, or other withdrawal criterion is met.
  Maintenance Therapy Comparator Arm: Phase 2 (every 21 days):
  Day 1: pemetrexed 500 mg/m^2
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Pemetrexed — Administered intravenously as a continuous 10-minute infusion
Drug: Cisplatin — Administered intravenously as a continuous 1-hour infusion
Drug: LY2603618 — Administered intravenously as a continuous 1-hour infusion
  Arms: Phase 1: LY2603618 130 to 275 mg; Phase 2: Pemetrexed + Cisplatin + LY2603618

SUMMARY:
LY2603618 is a selective inhibitor of the deoxyribonucleic acid (DNA) damage checkpoint kinase 1 (CHK1). It was being developed as a chemotherapeutic-enhancing agent in the treatment of cancer. Phase 1 studies have shown the feasibility of combining LY2603618 with either gemcitabine or pemetrexed. The objective of this study was to find the dose of LY2603618 that can be safely combined with standard doses of pemetrexed and cisplatin and to test if this triplet offered a significant improvement in progression-free survival (PFS) in participants with Stage IV nonsquamous non-small cell lung cancer (NSCLC) in the first-line of palliative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 portion:

  * Participants with a cytologic or histologic diagnosis of nonsquamous NSCLC that is classified as Stage IV according to the 7th edition of the American Joint Committee on Cancer (AJCC) classification and for whom the combination of pemetrexed and cisplatin is deemed to be appropriate
  * Participants with histologic or cytologic diagnosis of malignant mesothelioma that is unresectable
  * Participants with histologic or cytologic diagnoses of advanced or metastatic solid tumors who are not candidates for any standard therapy and for whom the combination with pemetrexed and cisplatin is deemed to be appropriate
* Phase 2 portion:

  * Have a histological diagnosis of NSCLC other than predominantly squamous cell histology that is classified as Stage IV according to the 7th edition of the AJCC classification
  * Eligible for a first line of palliative treatment with a platinum doublet
  * Have archived or fresh tumor tissue (not cytology)
* Phase 1 participants can have measurable or nonmeasurable disease. Phase 2 participants must have at least 1 measurable lesion according to Investigational New Drug (Response Evaluation Criteria in Solid Tumors [RECIST], v1.1) definitions. Tumor lesions located in a previously irradiated area can be considered measurable if they are new or if have shown unequivocal progression.
* Have a performance status ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have adequate hematologic, hepatic, and renal organ function
* Prior radiation therapy for treatment of cancer is allowed to <25% of the bone marrow, and participants must have recovered from the acute toxic effects of their treatment prior to study enrollment. Prior radiation to the whole pelvis is not allowed. Prior radiotherapy must be completed at least 4 weeks before study entry
* For women: Must be surgically sterile, postmenopausal, or compliant with a highly reliable contraceptive method (failure rate <1%) during and for 6 months after the treatment period; must have a negative serum or urine pregnancy test within 7 days before study enrollment and must not be breast-feeding. For men: Must be surgically sterile or compliant with a contraceptive regimen during and for 6 months after the treatment period

Exclusion Criteria:

* Have serious preexisting medical conditions or serious concomitant systemic disorders that would compromise the safety of the participant or his/her ability to complete the study, at the discretion of the investigator (for example, unstable angina pectoris or uncontrolled diabetes mellitus). Special attention should be paid to kidney and heart conditions that may be worsened with cisplatin treatment or hydration
* Have central nervous system (CNS) metastases (unless the participant has completed successful local therapy for CNS metastases and has been off corticosteroids for at least 4 weeks before starting study therapy). A screening computed tomography scan or magnetic resonance imaging before enrollment in the absence of a clinical suspicion of brain metastases is not required.
* Have current active infection that would, in the opinion of the investigator, compromise the participant's ability to tolerate therapy
* Have known allergy to pemetrexed, cisplatin, LY2603618, or any ingredient of pemetrexed, cisplatin, or LY2603618
* Have clinically significant (by physical exam) third-space fluid collections; for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry
* Participants taking non-steroidal anti-inflammatory drugs who cannot interrupt the treatment appropriately according to the guidelines
* Have received a recent yellow-fever vaccination (within 28 days of enrollment) or are receiving concurrent yellow-fever vaccination
* Phase 1 portion:

  * Have received more than 2 previous lines of chemotherapy for the advanced/metastatic disease
  * Have received more than 6 cycles of therapy containing an alkylating agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-02; Primary Completion 2013-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY(1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- Germany (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim, Baden-Wurttemberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster, Nordhein-Westfalen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coswig, Saxony
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Immenhausen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rheine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mataró, Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón, Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oviedo, Principality of Asturias
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Girona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville

REFERENCES:
- [Derived] Wehler T, Thomas M, Schumann C, Bosch-Barrera J, Vinolas Segarra N, Dickgreber NJ, Dalhoff K, Sebastian M, Corral Jaime J, Alonso M, Hynes SM, Lin J, Hurt K, Bence Lin A, Calvo E, Paz-Ares L. A randomized, phase 2 evaluation of the CHK1 inhibitor, LY2603618, administered in combination with pemetrexed and cisplatin in patients with advanced nonsquamous non-small cell lung cancer. Lung Cancer. 2017 Jun;108:212-216. doi: 10.1016/j.lungcan.2017.03.001. Epub 2017 Mar 6. PMID 28625637
- [Derived] Calvo E, Chen VJ, Marshall M, Ohnmacht U, Hynes SM, Kumm E, Diaz HB, Barnard D, Merzoug FF, Huber L, Kays L, Iversen P, Calles A, Voss B, Lin AB, Dickgreber N, Wehler T, Sebastian M. Preclinical analyses and phase I evaluation of LY2603618 administered in combination with pemetrexed and cisplatin in patients with advanced cancer. Invest New Drugs. 2014 Oct;32(5):955-68. doi: 10.1007/s10637-014-0114-5. Epub 2014 Jun 20. PMID 24942404

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Pemetrexed + Cisplatin + LY2603618: Cycles 1-2 (21-day cycle):
  Day 1: pemetrexed 500 milligrams per square meter (mg/m^2) + cisplatin 75 mg/m^2
  Day 2: LY2603618 130 to 275 milligrams (mg)
  After 2 cycles, participants may have continued on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion was met.
  Pemetrexed, cisplatin, and LY2603618 were administered intravenously (IV) over 10 minutes, 1 hour, and 1 hour, respectively.
- Phase 2: Pemetrexed + Cisplatin + LY2603618: Cycles 1-4 (21-day cycle):
  Before 25 Oct 2012:
  Day 1: pemetrexed 500 mg/m^2 + cisplatin 75 mg/m^2
  Day 2: LY2603618 dose determined from phase 1 (275 mg)
  After 25 Oct 2012:
  Day 1: pemetrexed 500 mg/m^2 + cisplatin 75 mg/m^2
  After 4 cycles, participants may have continued on maintenance therapy until disease progression, unacceptable toxicity, or other withdrawal criterion was met.
  Maintenance therapy (every 21 days):
  Before 25 Oct 2012:
  Day 1: pemetrexed 500 mg/m^2
  Day 2: LY2603618 dose determined from phase 1 (275 mg)
  After 25 Oct 2012:
  Day 1: pemetrexed 500 mg/m^2
  If, as of 25 Oct 2012, the participant was in maintenance therapy and randomized to the experimental arm, the participant was eligible to continue with pemetrexed/LY2603618 therapy if the investigator deemed it was in the participant's best interest and the participant consented.
  Pemetrexed, cisplatin, and LY2603618 were administered IV over 10 minutes, 1 hour, and 1 hour, respectively.
- Phase 2: Pemetrexed + Cisplatin: Cycles 1-4 (21-day cycle):
  Day 1: pemetrexed 500 mg/m^2 + cisplatin 75 mg/m^2
  After 4 cycles, participants may have continued on maintenance therapy until disease progression, unacceptable toxicity, or other withdrawal criterion was met.
  Maintenance therapy (every 21 days):
  Day 1: pemetrexed 500 mg/m^2
  Pemetrexed was administered IV over 10 minutes and cisplatin was administered IV over 1 hour.
Period: Overall Study
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Started | 14 | 39 | 23
Received at Least 1 Dose of Study Drug | 14 | 39 | 22
Completed | 13 | 26 | 17
Not Completed | 1 | 13 | 6
Not completed — Adverse Event | 0 | 6 | 2
Not completed — Protocol Violation | 0 | 5 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Physician Decision | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Phase 1: Pemetrexed + Cisplatin + LY2603618: Cycles 1-2 (21-day cycle):
  Day 1: pemetrexed 500 mg/m^2 + cisplatin 75 mg/m^2
  Day 2: LY2603618 130 to 275 mg
  After 2 cycles, participants may have continued on study drug until disease progression, unacceptable toxicity, or other withdrawal criterion was met.
  Pemetrexed, cisplatin, and LY2603618 were administered IV over 10 minutes, 1 hour, and 1 hour, respectively.
- Phase 2: Pemetrexed + Cisplatin: Cycles 1-4 (21-day cycle):
  Day 1: pemetrexed 500 mg/m^2 + cisplatin 75 mg/m^2
  After 4 cycles, participants may have continued on maintenance therapy until disease progression, unacceptable toxicity, or other withdrawal criterion was met.
  Maintenance therapy (every 21 days):
  Day 1: pemetrexed 500 mg/m^2
  Pemetrexed was administered IV over 10 minutes, and cisplatin was administered IV over 1 hour.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin | Total
Number analyzed (Participants) | 14 | 39 | 23 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.4) | 57.9 (10.1) | 56.4 (9.8) | 57.4 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 15 | 8 | 30
  Male | 7 | 24 | 15 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 39 | 23 | 76
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 7 | 24 | 12 | 43
  Germany | 7 | 15 | 11 | 33
Initial Pathological Diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma, Bronchiolalveolar | 0 | 0 | 1 | 1
  Adenocarcinoma, Colon | 1 | 0 | 0 | 1
  Adenocarcinoma, Lung | 8 | 38 | 19 | 65
  Adenocarcinoma, Moderately Diff., Lung | 0 | 0 | 1 | 1
  Carcinoma, Ampulla of Vater | 1 | 0 | 0 | 1
  Carcinoma, Breast | 1 | 0 | 0 | 1
  Carcinoma, Large Cell, Lung | 0 | 0 | 1 | 1
  Carcinoma, Lung | 0 | 1 | 0 | 1
  Carcinoma, Non-small Cell, Poorly Diff, Lung | 1 | 0 | 0 | 1
  Carcinoma, Pancreas | 1 | 0 | 0 | 1
  Mesothelioma, Malignum | 1 | 0 | 0 | 1
  Pleuritis Carcinomatosa | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death) as follows: 0 - Fully Active; 1 - Ambulatory, Restricted Strenuous Activity; 2 - Ambulatory, No Work Activities; 3 - Partially Confined to Bed, Limited Self Care; 4 - Completely Disabled; and 5 - Dead.
  Participants
    ECOG Status 0 | 11 | 9 | 7 | 27
    ECOG Status 1 | 3 | 30 | 15 | 48
    Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Progression-Free Survival Time
Description: Progression-free survival (PFS) time is defined as the time from the date of randomization to the first date of documented objective progressive disease (PD) or death from any cause. For participants who were not known to have had objective PD as of the data inclusion cut-off date for a particular analysis, PFS was censored at the date of the last objective progression-free disease assessments. For participants who took any subsequent systemic anticancer therapy prior to progression, PFS was censored at the date of the last objective progression-free disease assessment prior to the start date of any subsequent systemic anticancer therapy. PFS time was summarized using Kaplan-Meier estimates.
Time Frame: Randomization up to first date of PD or death from any cause (up to 6 months after the last participant entered treatment)
Population: All randomized Phase 2 participants.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Number analyzed (Participants) | 39 | 23
months | 4.7 [4.2 to 7.1] | 1.5 [1.3 to 2.9]
Statistical Analysis 1: Comparison: Phase 2: Pemetrexed + Cisplatin + LY2603618 vs Phase 2: Pemetrexed + Cisplatin; The analysis for comparing progression-free survival time between the treatment arms used a Bayesian Augmented Control model with a hierarchical random-effects distribution on treatment effects. The final model incorporated historical data from a completed Phase 3 study (NCT00789373) to augment the prospective control arm data; Test type: Superiority or Other; Bayesian Posterior Probability = 0.96 — Pemetrexed + cisplatin + LY2603618 was considered superior to pemetrexed + cisplatin if the posterior probability of superiority exceeded 0.85

2. Primary Outcome: Phase 1: Recommended Phase 2 Dose of LY2603618
Description: The recommended Phase 2 dose for LY2603618 when administered approximately 24 hours after pemetrexed and cisplatin was based on the maximum tolerated dose (MTD) and achievement of predefined LY2603618 plasma systemic exposures targets (area under the LY2603618 plasma concentration versus time curve from time zero to infinity [AUC(0-∞)] >21,000 nanogram*hour/milliliter [ng*h/mL] and maximum LY2603618 plasma concentration [Cmax] >2000 nanograms/milliliter [ng/mL]).
Time Frame: Time of first dose to last dose
Population: Phase 1 participants who received at least 1 dose of any of the study drugs.
Measure: Number; unit: mg
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618
Number analyzed (Participants) | 14
mg | 275

3. Secondary Outcome: Phase 2: Overall Survival
Description: Overall survival (OS) time is defined as the time from the date of randomization to the date of death from any cause. For participants not known to have died as of the data cut-off date, OS time was censored at the last contact date the participant was known to be alive prior to the data cut-off date. OS was summarized using Kaplan-Meier estimates.
Time Frame: Randomization to the date of death from any cause through the time of study discontinuation (approximately 12 months after last participant was randomized)
Population: All randomized Phase 2 participants.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Number analyzed (Participants) | 39 | 23
months | 12.9 [9.3 to NA] — The upper bound of the 90% confidence interval was not calculable. | 6.6 [4.2 to 19.4]
Statistical Analysis 1: Comparison: Phase 2: Pemetrexed + Cisplatin + LY2603618 vs Phase 2: Pemetrexed + Cisplatin; Test type: Superiority or Other; p = 0.2294, Log Rank — The test of treatment effect was conducted at a 2-sided alpha level of 0.10

4. Secondary Outcome: Phase 2: Overall Tumor Response Rate: Percentage of Participants Who Achieved a Confirmed Best Response of Completed Response (CR) or Partial Response (PR)
Description: Overall response rate is the best response of CR or PR as classified by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST, v1.1) guidelines. CR is defined as the disappearance of all target and non-target lesions, normalization of tumor marker level of non-target lesions, and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm). PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Randomization until date of disease progression (up to 6 months after the last participant was randomized)
Population: All randomized Phase 2 participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Number analyzed (Participants) | 39 | 23
percentage of participants | 43.6 [28.0 to 60.0] | 21.7 [7.0 to 44.0]
Statistical Analysis 1: Comparison: Phase 2: Pemetrexed + Cisplatin + LY2603618 vs Phase 2: Pemetrexed + Cisplatin; Test type: Superiority or Other; p = 0.0824, Chi-squared — The test of treatment effect was conducted at a 2-sided alpha level of 0.10

5. Secondary Outcome: Phase 2: Change in Tumor Size
Description: Change in tumor size was based on tumor measurements collected according to RECIST, v1.1 guidelines. Tumor size is the sum of the tumor measurements (longest diameters) of target lesions at each tumor evaluation. Change in tumor size was defined as the change in log tumor size from baseline evaluation to the evaluation at the end of Cycle 2.
Time Frame: Baseline, end of Cycle 2
Population: Participants with measureable disease (target lesions) at baseline who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Number analyzed (Participants) | 39 | 22
centimeters | -0.30 (0.541) | -0.14 (0.277)
Statistical Analysis 1: Comparison: Phase 2: Pemetrexed + Cisplatin + LY2603618 vs Phase 2: Pemetrexed + Cisplatin; Test type: Superiority or Other; p = 0.4924, Wilcoxon (Mann-Whitney) — The test of treatment effect was conducted at a 2-sided alpha level of 0.10

6. Secondary Outcome: Phase 1: Pharmacokinetic: Maximum Plasma Concentration (Cmax) (LY2603618)
Description: Cmax is reported for each LY2603618 dose level on Cycle 1 /Day 2 and Cycle 2 /Day 2. The number of pharmacokinetic observations (n) used in the analysis is presented for each dose level and time point.
Time Frame: Cycle 1/Day 2 - immediately prior to end of LY2603618 infusion, and 1, 3, 6, 24, 48, 72, and 144 hours postdose; Cycle 2/Day 2 - predose, immediately prior to end of LY2603618 infusion, and 1, 3, 6, 24, 48, 72, and 144 hours postdose
Population: Phase 1 participants who received at least 1 dose of LY2603618 and had samples collected for pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618
Number analyzed (Participants) | 13
ng/mL
  130 mg, Cycle 1/Day 2: number analyzed (Participants) | 3
  130 mg, Cycle 1/Day 2 | 1810 (14)
  130 mg, Cycle 2/Day 2: number analyzed (Participants) | 3
  130 mg, Cycle 2/Day 2 | 1730 (43)
  185 mg, Cycle 1/Day 2: number analyzed (Participants) | 3
  185 mg, Cycle 1/Day 2 | 2200 (33)
  185 mg, Cycle 2/Day 2: number analyzed (Participants) | 3
  185 mg, Cycle 2/Day 2 | 2190 (58)
  240 mg, Cycle 1/Day 2: number analyzed (Participants) | 3
  240 mg, Cycle 1/Day 2 | 3470 (27)
  240 mg, Cycle 2/Day 2: number analyzed (Participants) | 3
  240 mg, Cycle 2/Day 2 | 2750 (63)
  275 mg, Cycle 1/Day 2: number analyzed (Participants) | 3
  275 mg, Cycle 1/Day 2 | 4130 (29)
  275 mg, Cycle 2/Day 2: number analyzed (Participants) | 4
  275 mg, Cycle 2/Day 2 | 3620 (23)

7. Secondary Outcome: Phase 1: Pharmacokinetic: Cmax (Pemetrexed and Cisplatin)
Description: Cmax for pemetrexed and total platinum (t-platinum) from cisplatin is reported. The number of pharmacokinetic observations (n) used in the analysis is presented for each drug.
Time Frame: Pemetrexed: Cycle 1/Day 1 - immediately prior to end of pemetrexed infusion and 1, 2, 6 and 24 hours postdose. Cisplatin: Cycle 1/Day 1 - immediately prior to end of cisplatin infusion and 0.5, 1, 2, 6, 24, 72, 96, and 168 hours postdose.
Population: Phase 1 participants who received at least 1 dose of pemetrexed or cisplatin and had samples collected for pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618
Number analyzed (Participants) | 14
ng/mL
  Pemetrexed | 88300 (28)
  T-platinum from cisplatin | 3710 (43)

8. Secondary Outcome: Phase 1: Pharmacokinetic: Area Under the Plasma Concentration Versus Time Curve (AUC) (LY2603618)
Description: AUC from time zero to 24 hours (AUC[0-24]), AUC from time zero to the last time point with a measurable concentration (AUC[0-tlast]), and AUC from time zero to infinity (AUC[0-∞]) values are reported for each LY2603618 dose level on Cycle 1 /Day 2 and Cycle 2 /Day 2. The number of pharmacokinetic observations (n) used in the analysis is presented for each dose level and time point.
Time Frame: Cycle 1/Day 2 - immediately prior to end of LY2603618 infusion and 1, 3, 6, 24, 48, 72, and 144 hours postdose; Cycle 2/Day 2 - predose, immediately prior to end of LY2603618 infusion, and 1, 3, 6, 24, 48, 72, and 144 hours postdose
Population: Phase 1 participants who received at least 1 dose of LY2603618 and had samples collected for pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618
Number analyzed (Participants) | 13
ng*h/mL
  130 mg, Cycle 1/Day 2, AUC(0-24): number analyzed (Participants) | 3
  130 mg, Cycle 1/Day 2, AUC(0-24) | 8700 (30)
  130 mg, Cycle 2/Day 2, AUC(0-24): number analyzed (Participants) | 3
  130 mg, Cycle 2/Day 2, AUC(0-24) | 9780 (43)
  130 mg, Cycle 1/Day 2, AUC(0-tlast): number analyzed (Participants) | 3
  130 mg, Cycle 1/Day 2, AUC(0-tlast) | 10200 (26)
  130 mg, Cycle 2/Day 2, AUC(0-tlast): number analyzed (Participants) | 3
  130 mg, Cycle 2/Day 2, AUC(0-tlast) | 11300 (44)
  130 mg, Cycle 1/Day 2, AUC(0-∞): number analyzed (Participants) | 3
  130 mg, Cycle 1/Day 2, AUC(0-∞) | 10200 (26)
  130 mg, Cycle 2/Day 2, AUC(0-∞): number analyzed (Participants) | 3
  130 mg, Cycle 2/Day 2, AUC(0-∞) | 11300 (45)
  185 mg, Cycle 1/Day 2, AUC(0-24): number analyzed (Participants) | 3
  185 mg, Cycle 1/Day 2, AUC(0-24) | 13800 (119)
  185 mg, Cycle 2/Day 2, AUC(0-24): number analyzed (Participants) | 3
  185 mg, Cycle 2/Day 2, AUC(0-24) | 12500 (170)
  185 mg, Cycle 1/Day 2, AUC(0-tlast): number analyzed (Participants) | 3
  185 mg, Cycle 1/Day 2, AUC(0-tlast) | 18300 (192)
  185 mg, Cycle 2/Day 2, AUC(0-tlast): number analyzed (Participants) | 3
  185 mg, Cycle 2/Day 2, AUC(0-tlast) | 14800 (217)
  185 mg, Cycle 1/Day 2, AUC(0-∞): number analyzed (Participants) | 3
  185 mg, Cycle 1/Day 2, AUC(0-∞) | 18400 (193)
  185 mg, Cycle 2/Day 2, AUC(0-∞): number analyzed (Participants) | 3
  185 mg, Cycle 2/Day 2, AUC(0-∞) | 15700 (253)
  240 mg, Cycle 1/Day 2, AUC(0-24): number analyzed (Participants) | 3
  240 mg, Cycle 1/Day 2, AUC(0-24) | 26200 (19)
  240 mg, Cycle 2/Day 2, AUC(0-24): number analyzed (Participants) | 3
  240 mg, Cycle 2/Day 2, AUC(0-24) | 22100 (31)
  240 mg, Cycle 1/Day 2, AUC(0-tlast): number analyzed (Participants) | 3
  240 mg, Cycle 1/Day 2, AUC(0-tlast) | 32200 (21)
  240 mg, Cycle 2/Day 2, AUC(0-tlast): number analyzed (Participants) | 3
  240 mg, Cycle 2/Day 2, AUC(0-tlast) | 27300 (31)
  240 mg, Cycle 1/Day 2, AUC(0-∞): number analyzed (Participants) | 3
  240 mg, Cycle 1/Day 2, AUC(0-∞) | 32300 (21)
  240 mg, Cycle 2/Day 2, AUC(0-∞): number analyzed (Participants) | 3
  240 mg, Cycle 2/Day 2, AUC(0-∞) | 27500 (31)
  275 mg, Cycle 1/Day 2, AUC(0-24): number analyzed (Participants) | 4
  275 mg, Cycle 1/Day 2, AUC(0-24) | 28900 (24)
  275 mg, Cycle 2/Day 2, AUC(0-24): number analyzed (Participants) | 4
  275 mg, Cycle 2/Day 2, AUC(0-24) | 23500 (31)
  275 mg, Cycle 1/Day 2, AUC(0-tlast): number analyzed (Participants) | 4
  275 mg, Cycle 1/Day 2, AUC(0-tlast) | 38100 (36)
  275 mg, Cycle 2/Day 2, AUC(0-tlast): number analyzed (Participants) | 4
  275 mg, Cycle 2/Day 2, AUC(0-tlast) | 30800 (44)
  275 mg, Cycle 1/Day 2, AUC(0-∞): number analyzed (Participants) | 4
  275 mg, Cycle 1/Day 2, AUC(0-∞) | 38300 (37)
  275 mg, Cycle 2/Day 2, AUC(0-∞): number analyzed (Participants) | 4
  275 mg, Cycle 2/Day 2, AUC(0-∞) | 30900 (44)

9. Secondary Outcome: Phase 1: Pharmacokinetic: AUC (Pemetrexed and Cisplatin)
Description: AUC(0-tlast) and AUC(0-∞) values are reported for pemetrexed and t-platinum from cisplatin. The number of pharmacokinetic observations (n) used in the analysis is presented for each drug.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618
Number analyzed (Participants) | 14
ng*h/mL
  Pemetrexed, AUC(0-tlast) | 159000 (35)
  Pemetrexed, AUC (0-∞) | 160000 (35)
  T-platinum from cisplatin, AUC (0-tlast) | 163000 (26)
  T-platinum from cisplatin, AUC (0-∞) | 269000 (26)

10. Secondary Outcome: Phase 2: Pharmacokinetic: Cmax (LY2603618)
Time Frame: Cycle 1/Day 2 - predose, immediately prior to the end of the LY2603618 infusion, and 2-6, 24-48, and 72-96 hours postdose
Population: Phase 2 participants who received at least 1 dose of LY2603618 and had samples collected for pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 2: Pemetrexed + Cisplatin + LY2603618
Number analyzed (Participants) | 33
ng/mL | 4130 (66)

11. Secondary Outcome: Phase 2: Pharmacokinetic: AUC (LY2603618)
Description: AUC (0-24), AUC(0-tlast), and AUC(0-∞) values are reported for LY2603618. The number of pharmacokinetic observations (n) used in the analysis is presented.
Time Frame: as for outcome 10
Population: Phase 2 participants who received at least 1 dose of LY2603618 and had samples collected for pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 2: Pemetrexed + Cisplatin + LY2603618
Number analyzed (Participants) | 33
ng*h/mL
  AUC (0-24): number analyzed (Participants) | 32
  AUC (0-24) | 31400 (49)
  AUC (0-tlast): number analyzed (Participants) | 32
  AUC (0-tlast) | 39300 (58)
  AUC (0-∞): number analyzed (Participants) | 31
  AUC (0-∞) | 41100 (59)

12. Secondary Outcome: Phase 2: Change From Baseline to Long-term Follow up in Lung Cancer Symptom Scale (LCSS)
Description: Health-related quality of life and participant symptoms were assessed using the LCSS (patient scale). However, improper implementation of questionnaires at the site level reduced the sponsor's ability to accurately evaluate the impacted data. Therefore, the LCSS data should be interpreted with caution.
  The LCSS is a 9-item questionnaire. Six questions are symptom-specific measures for lung cancer (appetite, fatigue, cough, dyspnea, hemoptysis, and pain), and 3 summation items describe total symptomatic distress, activity status, and overall quality of life. Participant responses were measured using visual analogue scales (VAS) with 100-milliliter (mm) lines. Scores range from 0 (for best outcome) to 100 (for worst outcome). The Average Symptom Burden Index (ASBI) was calculated as the mean of 6 symptom-specific questions from the LCSS. The total LCSS score was calculated as the mean of 9 questions from the LCSS.
Time Frame: Randomization to the end of study (approximately 12 months after the last participant entered treatment)
Population: All enrolled Phase 2 participants who had the baseline LCSS assessment and at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Number analyzed (Participants) | 36 | 22
units on a scale
  Total LCSS: number analyzed (Participants) | 32 | 21
  Total LCSS | -10.7 (14.1) | -11.7 (15.1)
  ASBI: number analyzed (Participants) | 34 | 21
  ASBI | -11.6 (13.9) | -12.6 (15.4)

13. Secondary Outcome: Phase 1: Document Any Antitumor Activity Per Radiological Scans and/or Tumor Markers
Description: Overall response rate is presented. Overall response rate is defined as the percentage of participants with a best response of CR or PR as classified by the investigators according to RECIST, v1.1 criteria. CR is defined as the disappearance of all target and non-target lesions, normalization of tumor marker level of non-target lesions, and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Baseline through end of Phase 1
Population: All randomized Phase 1 participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618
Number analyzed (Participants) | 14
percentage of participants
  130 mg: number analyzed (Participants) | 3
  130 mg | 0 [0 to 0]
  185 mg: number analyzed (Participants) | 3
  185 mg | 66.7 [9.0 to 99.0]
  240 mg: number analyzed (Participants) | 4
  240 mg | 25.0 [1.0 to 81.0]
  275 mg: number analyzed (Participants) | 4
  275 mg | 0 [0 to 0]

14. Other Pre Specified Outcome: Deaths
Description: Deaths that occurred during the study are presented. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Randomization through 12 months after the last participant was randomized
Population: All enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Number analyzed (Participants) | 14 | 39 | 23
Participants
  Total deaths | 0 | 21 | 15
  Deaths while on treatment | 0 | 3 | 1
  Death within 30 days of last dose of study drug | 0 | 1 | 0
  Deaths during follow-up period | 0 | 17 | 14

15. Secondary Outcome: Phase 2: Proportion of Participants Receiving Maintenance Therapy
Time Frame: Cycle 5
Population: Zero participants analyzed. Treatment with LY2603618 was discontinued after 25 October 2012, data was not collected for analysis of the Phase 2: Proportion of Participants Receiving Maintenance Therapy.
Arm/Group | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Phase 2: Clinical Benefit Rate: Percentage of Participant Who Achieved a Response of Stable Disease (SD), Partial Response (PR), or Complete Response (CR)
Description: Clinical benefit rate is the best response CR, PR, or SD as classified by the investigators according to the RECIST, v1.1 guidelines. CR is defined as the disappearance of all target and non-target lesions, normalization of tumor marker level of non-target lesions, and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameter since treatment started. Clinical benefit rate is calculated as a total number of participants with CR, PR, or SD divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Randomization until date of disease progression or death (up to 6 months after the last participant was randomized)
Population: All randomized Phase 2 participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Number analyzed (Participants) | 39 | 23
percentage of participants | 69.2 [52.0 to 83.0] | 47.8 [27.0 to 69.0]
Statistical Analysis 1: Comparison: Phase 2: Pemetrexed + Cisplatin + LY2603618 vs Phase 2: Pemetrexed + Cisplatin; Test type: Superiority or Other; p = 0.0946, Chi-squared — The test of treatment effect was conducted at a 2-sided alpha level of 0.10

ADVERSE EVENTS:
Arm/Group | Phase 1: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin + LY2603618 | Phase 2: Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 1/14 | 16/39 | 6/22
Other Adverse Events (participants affected / at risk) | 14/14 | 37/39 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Pemetrexed + Cisplatin + LY2603618 (N=14) | Phase 2: Pemetrexed + Cisplatin + LY2603618 (N=39) | Phase 2: Pemetrexed + Cisplatin (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1: Pemetrexed + Cisplatin + LY2603618 (N=14) | Phase 2: Pemetrexed + Cisplatin + LY2603618 (N=39) | Phase 2: Pemetrexed + Cisplatin (N=22)
Anaemia (Blood and lymphatic system disorders) | 3 (16) | 7 (16) | 3 (6)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 5 (11) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (13) | 8 (11) | 4 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (10) | 1 (1) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Ototoxicity (Ear and labyrinth disorders) | 0 (0) | 8 (22) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (4) | 5 (7) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 3 (4) | 2 (3) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (9) | 2 (3) | 3 (4)
Eye oedema (Eye disorders) | 0 (0) | 3 (4) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Papilloedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (4) | 18 (30) | 8 (13)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 11 (17) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (44) | 30 (106) | 15 (27)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (13) | 18 (42) | 6 (9)
Asthenia (General disorders) | 2 (2) | 17 (82) | 5 (12)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (2)
Chest pain (General disorders) | 0 (0) | 4 (4) | 2 (3)
Chills (General disorders) | 1 (2) | 1 (2) | 3 (4)
Fatigue (General disorders) | 13 (35) | 14 (23) | 14 (21)
Infusion site extravasation (General disorders) | 0 (0) | 2 (2) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 10 (22) | 4 (7)
Oedema (General disorders) | 3 (3) | 4 (7) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 6 (10) | 3 (3)
Pyrexia (General disorders) | 6 (8) | 10 (19) | 9 (10)
Hypersensitivity (Immune system disorders) | 1 (3) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5) | 2 (2)
Paronychia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (5) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Blood creatinine increased (Investigations) | 1 (3) | 3 (5) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 4 (4) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (6) | 3 (4) | 2 (5)
Platelet count decreased (Investigations) | 1 (3) | 2 (8) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 3 (4) | 2 (3)
White blood cell count decreased (Investigations) | 1 (4) | 1 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 14 (45) | 12 (19)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (11) | 4 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 6 (12) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (2) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (5) | 8 (17) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3)
Neurotoxicity (Nervous system disorders) | 0 (0) | 7 (9) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (5) | 4 (4) | 1 (1)
Paresis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 2 (2)
Depression (Psychiatric disorders) | 1 (2) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (6) | 4 (5) | 3 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0/7 (0) | 1/15 (1) | 0/8 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 8 (19) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (16) | 7 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (5) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4) | 2 (2)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Catheterisation venous (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 3 (7) | 3 (4) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment was halted on 25 October 2012 due to a numerical imbalance in events of thromboembolic nature between the experimental arm and the control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days